CLINICAL TRIAL: NCT06485050
Title: Photodynamic Therapy as Adjuvant Therapy to Topical Antifungal Treatments for Onychomycosis in Patients With Diabetes. A Prospective Case Series.
Brief Title: Photodynamic Therapy and Topical Antifungal for Onychomycosis in Patients With Diabetes.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, Jose Luis Lazaro Martinez, Head of the Diabetic foot Unit, Universidad Complutense de Madrid
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24/241-E
Record Dates: First submitted 2024-05-22; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Dermatologic Disease; Onychomycosis of Toenail; Diabetic Foot; Diabetes Mellitus
MeSH Terms: conditions — Skin Diseases; Diabetic Foot; Diabetes Mellitus | interventions — Photochemotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Photodynamic therapy with ciclopirox 8% (Experimental)
  Interventions: Combination Product: Photodynamic therapy

INTERVENTIONS:
Combination Product: Photodynamic therapy — Application of red laser-photodynamic therapy using "Rapid Podia" Laser diode® (MEDENCY). The following protocol will be followed: 1) mechanical debridement of the nail, 2) disinfection of the nail with alcohol, 3) application of topical photosensitiser (Toluidine blue gel) for 5 minutes with the area covered, 5) application of 635 nm diode laser for 10 minutes.
  Daily application of ciclopirox 8% with ethyl acetate, ethanol (96%), ketosteryl alcohol, hydroxypropyl chitosan and purified water.

SUMMARY:
There are different therapeutic alternatives for onychomycosis. Systemic therapy is widely used due to its easy accessibility, low cost and high efficacy, but may be associated with systemic adverse events and drug-drug interactions, so its use in patients with diabetes, immunocompromised and frequently take more than five drugs is not recommended even though these individuals are at serious risk of fungal infection. On the other hand, laser therapy would be contraindicated in patients with neuropathy or peripheral vascular disease (diabetic foot patients) because of possible burns. Topical antifungals or lacquers are associated with a low risk of systemic adverse events and drug-drug interactions and would therefore be the most appropriate treatment for patients with diabetic foot. However, they require very long treatment periods, are generally applied daily for 12 months to allow the normal nail to grow and replace the regions damaged by the infection and have a lower cure rate.

Because of all the above difficulties, there is a need to augment topical treatments in routine clinical practice with adjunctive therapies such as photodynamic therapy for the treatment of onychomycosis in patients with diabetes.

The main aim of this study is to observe the effectiveness and safety of the combination of photodynamic therapy with the usual antifungal treatment in consultation in patients with diabetes. Secondary aims have been defined as follows:

To determine whether 3 sessions of photodynamic therapy combined with topical therapy, over a period of 6 months, is sufficient to achieve clinical, mycological and complete cure of onychomycosis; And to analyse the influence of the type of onychomycosis (ODL, total dystrophic, superficial), the causal fungal agent (dermatophyte, mould or yeast) and the degree of severity of onychomycosis (through the OSI) on the response to treatment.

Patients included in the study will be visited every 2 weeks during the first two months, applying photodynamic therapy during visits 2, 3 and 4. Subsequently, a check-up will be performed two weeks after the last application of photodynamic therapy and monthly visits for the remainder of the study. At each visit and at subsequent check-ups, the nail plate and peri- and subungual hyperkeratotic tissue will be debrided and reamed in order to improve the effects of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diabetes diagnosed with toenail onychomycosis with positive microbiological culture/PCR.

Patients over 18 years of age.

Exclusion Criteria:

* Patients who have received topical or systemic antifungal treatment in the previous month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-04-17 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Main outcome | 6 months
  Number of participants with treatment-related adverse events as assessed by the effectiveness of the combination of photodynamic therapy with the usual antifungal treatment in the clinic in patients with diabetes, change from baseline in score on the Onychomycosis Severity Index (OSI), microbiological culture and polymerase chain reaction (PCR) at 6 months.

SECONDARY OUTCOMES:
Secondary outcome | 6 months
  Number of patients who are successfully cured with 3 sessions of photodynamic therapy combined with topical therapy, over a period of 6 months, is sufficient to achieve clinical, mycological and complete cure of onychomycosis with microbiological culture and PCR results.
Secondary outcome | 6 months
  Influence of the type of onychomycosis (ODL, total dystrophic, superficial) and the degree of severity of onychomycosis by the OSI score on the response to treatment at 6 months.
Secondary outcome | 6 months
  Influence of the causal fungal agent (dermatophyte, mould or yeast) and the degree of severity of onychomycosis by the OSI score on the response to treatment at 6 months.

CONTACTS AND LOCATIONS:
Locations (1):
- University podiatry clinic (Complutense University of Madrid), Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes